CLINICAL TRIAL: NCT06232473
Title: Efficacy of Patient Education and Duloxetine, Alone or in Combination, for Patients With Multisystem Functional Somatic Disorder
Brief Title: Patient Education and Duloxetine, Alone and in Combination, for Patients With Multisystem Functional Somatic Disorder
Acronym: EDULOX
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: Central Denmark Region (Other); University of Aarhus (Other); Vejle Hospital (Other); Aalborg University Hospital (Other); TrygFonden, Denmark (Industry); Independent Research Fund Denmark (Industry)
Responsible Party: Sponsor
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9515
Record Dates: First submitted 2024-01-02; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Functional Disorder
Keywords: Patient Education; Duloxetine; Medically Unexplained Symptoms; SNRI; Bodily Distress Syndrome; Functional Somatic Symptoms; Functional Somatic Disorders; Randomized Controlled Trial; Biobank; Biomarker
MeSH Terms: conditions — Medically Unexplained Symptoms | interventions — Patient Education as Topic; Duloxetine Hydrochloride; Serotonin and Noradrenaline Reuptake Inhibitors; Benztropine

STUDY DESIGN:
Intervention Model Description: This is a nested design. The parent trial (EDULOX 1) is an open-labelled randomized controlled trial comparing patient education (PE) with enhanced usual care (EUC). The parent trial nests a concomitantly running, two-by-two factorial, double-blinded, randomised controlled trial (EDULOX 2) comparing duloxetine with active placebo in combination with the PE program or EUC.
  Participants in the parent trial will be randomized (open-label) to receive either EUC or the PE program. Participants in the nested trial will be randomized (open-label + blinded) to receive either EUC or PE along with either duloxetine or active placebo. This will result in a total of six randomization groups for the full EDULOX trial.
  A total of 424 participants will be recruited for the EDULOX parent trial, of these 212 participants will participate in the nested study drug trial.
  Biological material for the biobank will be collected from all participants and an additional 75 healthy controls.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization for both the open-label parent trial and the nested blinded study drug trial will be carried out using REDCap. The randomization code will be generated by an independent employee through REDCap. Coded (numbered) packs of study drug and active placebo will be produced according to the randomization schedule. Patients, clinicians, investigators, and all other staff involved in the conduct or data analysis of the nested trial will be masked to study drug treatment allocation for the duration of the study and throughout all data analysis. Patients and clinicians will be asked to guess allocated treatment (duloxetine or active placebo) and indicate reason at endpoints to evaluate blinding efficacy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Patient Education (Experimental): The patient education program consists of three individual sessions (consultations with the participant's doctor, one to one and a half hour duration each) and one group session (three hours in groups of up to 16 participants). The program focuses on providing patients with a positive and evidence-based understanding of their illness by providing an individualized bio-psycho-social explanation of multisystem functional somatic disorder.
  Interventions: Behavioral: Patient Education
- Enhanced Usual Care (Active Comparator): Inclusion consultation and final visit at end of treatment (week 12) are the only contacts provided to participants randomized to receive enhanced usual care.
  Interventions: Behavioral: Enhanced usual care
- Duloxetine and Enhanced Usual Care (Experimental): Duloxetine will be given as capsules orally once daily. Participants will commence with 2 weeks of 30 mg duloxetine and then increase the dose to 60 mg duloxetine (two capsules). If participants are unable to increase in dose due to adverse events, but still tolerate the initial dose of 30 mg duloxetine, this dose is kept for the remaining part of the trial. Treatment will continue for 8 weeks on highest dosis until primary endpoint (end of treatment). The dose is then reduced to 30 mg duloxetine for 1 week after which the study drug is discontinued.
  In addition, participants will recieve enhanced usual care as described above.
  Interventions: Drug: Duloxetine; Behavioral: Enhanced usual care
- Placebo and Enhanced Usual Care (Placebo Comparator): Participants will recieve the active placebo benztropine mesylate 0,5 mg. In order to best mimic the dosage increase of the duloxetine treatment program a passive placebo RAP will be added for the 8 weeks of high dosage treatment. Benztropine mesylate and passive placebo will be given as capsules orally, and will be re-encapsulated by the hospital pharmacy to assure identical appearance to the duloxetine capsules. Participants will commence with 2 weeks of 0.5 mg benztropine mesylate (one capsule) and continue with 0.5 mg benztropine mesylate and passive placebo RAP (two capsules) for 8 weeks. This will be end of treatment. Participants will then be asked to reduce to one capsule (0.5 mg benztropine mesylate) for 1 week after which the study drug is discontinued.
  In addition, participants will recieve enhanced usual care as decribed above.
  Interventions: Drug: Benztropine Mesylate 0.5 MG and passive placebo RAP; Behavioral: Enhanced usual care
- Patient Education and Duloxetine (Experimental): Participants in this arm will recieve patient education as described above. In addition, participants will recieve duloxetine as described above.
  Interventions: Behavioral: Patient Education; Drug: Duloxetine
- Patient Education and Placebo (Experimental): Participants in this arm will recieve patient education as described above. In addition, participants will recieve the placebo treatment as described above.
  Interventions: Behavioral: Patient Education; Drug: Benztropine Mesylate 0.5 MG and passive placebo RAP

INTERVENTIONS:
Behavioral: Patient Education — Please see arm desciption
  Arms: Patient Education; Patient Education and Duloxetine; Patient Education and Placebo
Drug: Duloxetine — Please see arm description
  Other Names: Cymbalta; SNRI
  Arms: Duloxetine and Enhanced Usual Care; Patient Education and Duloxetine
Drug: Benztropine Mesylate 0.5 MG and passive placebo RAP — Please see arm description
  Arms: Patient Education and Placebo; Placebo and Enhanced Usual Care
Behavioral: Enhanced usual care — Please see arm description
  Arms: Duloxetine and Enhanced Usual Care; Enhanced Usual Care; Placebo and Enhanced Usual Care

SUMMARY:
The goal of this clinical trial is to test if patient education or duloxetine can be used to treat multisystem functional somatic disorder (FSD). The main questions it aims to answer are:

* Does duloxetine work better than placebo in the treatment of FSD?
* Does patient education work better than usual treatment for FSD?
* Does the combination of patient education and duloxetine work better than using only one of these treatments?

Participants are patients with FSD. They will receive one of six different treatment combinations:

1. Patient education alone (three individual consultations with a doctor and one group session)
2. Treatment as usual (receiving the diagnosis and a short presentation of what FSD is)
3. Duloxetine
4. Active placebo (a treatment that looks like duloxetine and has similar side effects, but no known effect on FSD)
5. Patient education and duloxetine
6. Patient education and active placebo

Researchers will compare the groups receiving patient education with those receiving only treatment as usual to see if patient education is a better treatment than just receiving a diagnosis and short explanation. Furthermore, researchers will compare the groups receiving duloxetine to those receiving placebo to see if duloxetine works better than placebo. Finally, researchers will compare the groups receiving both patient education and duloxetine to those receiving only one of these treatments to see if the combination works better than the treatments given alone.

The researchers will also collect samples of blood and stool in a biobank to be used in future research.

DETAILED DESCRIPTION:
Background Functional somatic disorders (FSD) are characterized by specific patterns of persistent physical symptoms with a complex etiology involving a multiform interplay between physiological, psychological, and socio-cultural factors. Patients with FSD are prevalent in all medical settings and receive diagnoses such as fibromyalgia, chronic fatigue syndrome, irritable bowel syndrome, and other functional somatic syndromes (FSS) depending on which medical specialty they consult. Multisystem FSD describes a severely affected subgroup of patients who suffer from symptoms from multiple organ systems. The diagnosis can be operationalized by the criteria for the unifying research diagnosis bodily distress syndrome (BDS).

Multisystem FSD affects 1.3-2.2% of the general population. The condition inflicts suffering and is associated with a substantial socioeconomic impact, involving costly diagnostic examinations and procedures, sick leaves, and long-term disability.

Evidence on treatment options for multisystem FSD is emerging but not yet sufficient. A number of clinical trials investigating non-pharmacological interventions are available and clinical guidelines in some FSS, e.g. fibromyalgia and chronic primary pain, highlight the importance of patient education (PE). PE may support the effect of other treatments by empowering and engaging patients in managing their condition. As a stand-alone treatment, the effect of PE has only sparsely been investigated, yet a PE program targeting multisystem FSD has been tested in an uncontrolled pilot study with promising results.

Pharmacotherapy in FSS includes centrally acting drugs, especially antidepressants. In multisystem FSD, evidence exists for treatment with low-dose tricyclic antidepressants (TCA). Unfortunately, TCAs given in higher, antidepressive doses significantly reduces tolerability and thereby treatment potential for comorbid depression or anxiety which are common in multisystem FSD. Duloxetine, a serotonin-norepinephrine reuptake inhibitor (SNRI), offers effect sizes similar to low-dose TCA in FSS with a more favorable adverse event profile. Evidence furthermore suggests an effect on cognitive functioning. In addition to reducing symptoms in multisystem FSD, duloxetine could improve cognitive functioning and, if relevant, treat comorbid anxiety and depression.

From a clinical perspective, a synergic effect between a PE program and pharmacological treatment could be hypothesized. On one hand, PE may improve the effect of pharmacological treatment by balancing treatment expectations and enhancing treatment adherence. Conversely, pharmacological treatment may indirectly enhance the effect of PE by improving cognitive functioning and thereby improving the patients' ability to receive and implement relevant educational elements.

As mentioned above, the etiology of FSD is complex and especially the role of biological factors remains largely undiscovered. Research findings support involvement of the immune system, neuroendocrine and neurotransmitter systems, pain processing and gut microbiota. In order to investigate the relevance of such components in multisystem FSD, this study will collect blood, plasma and feces from participants and healthy controls in order to establish a biobank enabling future research in these relevant factors.

Purpose and aim The EDULOX trial aims to investigate the effect of a PE program compared with enhanced usual care (EUC) for patients with multisystem FSD in EDULOX1. Additionally, the study investigates the effect of treatment with duloxetine 60 mg daily against active placebo and explores the effect of combinations of the two interventions in EDULOX2. This is to our knowledge the first study to investigate the combination of medical treatment and PE for patients with multisystem FSD.

By establishing a biobank with blood, plasma and feces from both EDULOX participants and healthy controls, the EDULOX trial furthermore aims to identify possible biomarkers in multisystem FSD and relate these to the outcome measures in the study.

Hypothesis EDULOX1:

The primary hypothesis is that the PE program is superior to EUC in improving patient-rated health-related quality of life measured by a Short-Form Health Survey (SF-36) aggregate score and patient-rated overall health measured by the Clinical Global Improvement Scale (CGI).

Hypothesis EDULOX2:

The primary hypothesis is that duloxetine is superior to active placebo in improving the SF-36 aggregate score, the CGI and cognitive functioning measured by Cognitive Failures Questionnaire (CFQ) at end of treatment.

Exploratory hypothesis:

There is a synergistic effect of receiving both PE and duloxetine, i.e. participants receiving both interventions show larger improvement in SF-36 aggregate score and CGI, than would be expected from simple additive effect of each intervention.

Hypothesis biobank We hypothesize that the immune system, hypothalamic-pituitary-adrenal axis, neurotransmitter levels, symptom- and/or pain processes are changed, and that the gut microbiota is disturbed. Changes are correlated to the severity of symptoms.

Methods For study design please see separate segment in the clinical trial registration.

Setting The project is initiated and managed by the Research Clinic for Functional Disorders and Psychosomatics (RCF), Aarhus University Hospital (AUH), Denmark. Participants will be recruited from eligible patients from the RCF, AUH or patients referred to the RCF for possible participation from the Pain and Headache Clinic, AUH, Center for Functional Disorders, the Hospital Lillebælt, and the Center for Functional Disorders, Aalborg University Hospital.

Interventions Please see Arms and Interventions segment of the clinical trial registration.

Data sources and effect measures Data sources include patient-rated outcomes, clinician-rated outcomes, and a qualitative evaluation consisting of 10-15 patient interviews examining acceptability and patient experiences regarding the PE intervention.

Questionnaire data will be collected at 5 time points:

* T0: Baseline (before inclusion)
* T1: Week 0 (before randomization)
* T2: Week 6 (during treatment)
* T3: Week 12 (end of treatment, primary endpoint)
* T4: 3-months follow-up after end of treatment

Naturalistic follow-up measurements are collected at 12 and 24 months from randomization (T5 and T6).

Please see further details in the Outcome Measures segment of the clinical trial registration.

Acceptability and feasibility measures Acceptability and feasibility measures will be collected from the first 40 participants. Reasons for non-participation, drop-out and breaking protocol will be analyzed. These data will be used to identify any major obstacles for the smooth running of the EDULOX. Patient acceptancy will be investigated through the Experience of Service Questionnaire and through a qualitative interview study with 10-15 planned semi-structured interviews.

Feasibility criteria are based on prior studies and will include:

* Inclusion rate more than 85% on the PE trial and 45% on the duloxetine trial.
* Drop-out will be less than 15% (reasons for drop out will be analyzed)
* More than 90% of the participants allocated to receive PE completes the PE program by attending at least two individual sessions and the group PE session
* Missing data will be less than 15%
* Questionnaire response-rate of minimum 90% at baseline and minimum 85% for the endpoint questionnaires (12 weeks, T3)
* PE will prove acceptable to patients with a patient satisfaction score of moderate to high
* Blinding in the duloxetine trial will be sufficient

Safety and monitoring The safety profile of duloxetine is well-described for patients with fibromyalgia and patients will be informed about the most common and the most severe adverse events for both duloxetine and benztropine mesylate.

Safety is assessed by collecting information on adverse events by the clinician (final visit, all contacts regarding adverse events). Patients are instructed to contact the project nurse by phone if experiencing any problems with the study drug. The nurse will have access to advice from medical doctors. Project workers can be contacted by telephone at all times if acute unblinding is required.

The project will be conducted in accordance with the Helsinki Declaration (II). General procedures for quality control and quality assurance will be followed. All protocol violations will be recorded. The quality and safety of the project are monitored by the Good Clinical Practise GCP unit at Department of Clinical Medicine, Aarhus University.

Discussion Solid and rigidly designed intervention studies for patients suffering from severe functional somatic disorders are highly needed. A documented positive effect of duloxetine will provide clinicians with an easily delivered pharmacological treatment option, and furthermore, new cost-effective treatment approaches arise if study results suggest a synergic effect of the combination of duloxetine and PE.

Such results could support the development of a stepped care model securing better treatment faster for those who can benefit from treatment in less specialized settings. This is of great significance since many clinics currently have waiting lists of more than a year, risking possible chronification of symptoms while patients wait for relevant treatment.

A biobank with relevant biological samples may enable future research into important etiological factors of FSD which remains largely uncovered. Insight into such possible biomarkers and their relation to the severity of the disorder could open up new possibilities for targeted treatment.

ELIGIBILITY:
Inclusion criteria for the parent trial:

* A diagnosis of multisystem functional somatic disorder (operationalized as fulfilling the criteria for the research diagnosis multiorgan bodily distress syndrome)
* Symptoms present for at least six months at the time of inclusion
* Multisystem functional somatic disorder is the predominant health complaint, i.e. concurrent physical or psychiatric illness is stable and well controlled and symptoms can be separated from BDS symptoms
* Understands and speaks Danish fluently and is able to follow and benefit from an educational program
* First-time referral to specialized treatment for functional somatic disorder

Additional inclusion criteria for the nested study drug trial:

* Use of efficient contraception for women in the fertile age (contractive pills, intrauterine device, deposit injections of gestagen, subdermal implant, hormone vaginal ring, or transdermal deposit plaster)
* Men with a pregnant or non-pregnant female partner in the fertile age must use a condom in the full length of the trial plus a minimum of one week after end of study drug treatment

Exclusion criteria for parent trial:

* Participation in psychotherapy or educational programs specifically for FSD within the past 12 months
* Current or previous diagnosis of mania, bipolar disorder, psychosis, severe agitation, imminent deliria or psychotic symptoms
* SCAN or clinical diagnosis of moderate to severe depression, anxiety or other psychiatric disorders
* Current affective disorder requiring fast initiation or continuation of psychiatric pharmacological treatment or psychiatric monitoring
* Alcohol, substance or medicine abuse or addiction

Additional exclusion criteria for the nested trial

* Treatment with duloxetine for a period of at least 8 successive weeks within the past 6 months
* Allergy to study medication or excipients in study medication
* Serious or unstabile somatic illness, e.g. stroke, Alzheimers disease, ischemic heart disease, epilepsy, fructose intolerance, glucosegalactose malabsorption, invertase-isomaltase insufficiency, increased intraocular pressure, uncontrolled narrow-angle glaucoma, hemodialysis, hemophilia, reduced platelet function, increased bleeding tendency, Raynaud's phenomenon, uncontrolled hypertension, prostate hypertrophy, urin retension or previous anaphylactic shock
* Severe renal impairment with creatinine clearance <30 ml / min. (risk of increased plasma concentration of duloxetine)
* Liver disease with reduced function with affected blood tests (risk of increased plasma concentration of duloxetine)
* Sweat gland disorder (risk of hyperthermia in high temperatures related to use of benztropine)
* Current pregnancy or lactation
* Concomitant use of CNS-acting drugs (drugs with pain-modulating or antidepressant properties and others) besides paracetamol and ibuprofen (escape medication in restricted doses). When clinically relevant and safe, the prohibited medication is gradually titrated down at the time of study inclusion, and treatments are discontinued at least 2 weeks before the study drug treatment begins)
* Concomitant use of drugs interacting with or contraindicating duloxetine treatment, e.g. serotonergic antidepressants (SSRI og TCA præparater, e.g. clomipramine or amitriptyline), dietary supplement St. John's wort (Hypericum perforatum), venlafaxine, MAO inhibitants or triptanes, tramadol, pethidin and tryptophan (risik of serotonin syndrome)
* Concomitant use of potent CYP1A2-inhibitants, e.g. fluvoxamine, ciprofloxacine og enoxacine (risk of increased plasma concentration of duloxetine)
* Concomitant use of non-selective, irreversible or selective, reversible monoaminoxidase (MAO) inhibitants; at least 14 days between termination of treatment with MAO-inhibitants and beginning of treatment with duloxetine. Additionally, treatment with MAO-inhibitants are not allowed before duloxetine treatment has been terminated for 5 days (risk of serotonin syndrome)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 424 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
Mean difference between groups in Short-Form Health Survey (SF-36) aggregate score | T0 (baseline, before assessment), T1(after inclusion, before randomization), T2 (week 6, mid-treatment), T3 (primary endpoint, week 12), T4 (3-month after end of treatment), T5 (1-year follow-up), T6 (2-year follow-up)
  Patient-rated health-related quality of life is measured by an aggregate score of the SF-36 subscales "physical functioning", "bodily pain" and "vitality" at endpoint (week 12).
  Minimum score is 15 and maximum score is 62 with lower scores indicating worse health related quality of life. Primary outcome will be measured as the change from baseline to primary endpoint (12 weeks), but data will be collected on several timepoints to describe the development on the score
Mean difference between groups in Clinical Global Improvement Scale (CGI) score | T3 (primary endpoint, 12 weeks), T4 (3-month follow-up), T5 (1-year follow-up), T6 (2-year follow-up)
  Patient-rated overall health improvement measured by the 5-point CGI. General health is rated as "much worse", "worse", "unchanged", "better" or "much better" in response to the question: "How do you consider your health status now compared with when you first came to the clinic?".

SECONDARY OUTCOMES:
Mean difference between groups in the Symptom Checklist (SCL-92) score on subscales somatic symptoms (SCL-som), anxiety and depression (SCL-anx 4, SCL-depr 6) | T0 (baseline, before assessment), T1(before randomization), T2 (week 6, mid-treatment), T3 (primary endpoint, 12 weeks), T4 (3-month follow-up), T5 (1-year follow-up), T6 (2-year follow-up)
  Health related physical and psychological functioning will be measured using relevant subscales of the Somatisation score measured using the SCL-92.
  SCL-som contains 12 items, SCL-anx 4 and SCL-depr 6 contains a total of 10 items. All items are scored on a 5 point Likert scale. Higher scores indicates more symptoms.
Mean difference between groups in the Bodily Distress Syndrome (BDS) check-list score | T0 (baseline, before assessment), T1(before randomization), T3 (primary endpoint, 12 weeks), T4 (3-month follow-up), T5 (1-year follow-up), T6 (2-year follow-up)
  The BDS check-list will be used to measure the severity of FSD symptoms. The BDS symptom score ranges from 0-100, with each of the 25 symptoms being scored on a Likert scale from 0-4. A higher score indicates more symptoms.
Mean difference between groups in Cognitive Failures Questionnaire (CFQ) score | T1(before randomization), T2 (week 6, mid-treatment), T3 (primary endpoint, 12 weeks)
  Cognitive functioning will be measured using the 25 item CFQ. The total score ranges from 0-100 with a higher score indicating a more impaired cognitive functioning.
Mean difference between groups in Whiteley-6-R score | T0 (baseline, before assessment), T1(before randomization), T2 (week 6, mid-treatment), T3 (primary endpoint, 12 weeks), T4 (3-month follow-up), T5 (1-year follow-up), T6 (2-year follow-up)
  Whiteley-6-R is used to measure illness worry. This 6 item score ranges from 0-24 with a higher score indicating more illness worry.
Mean difference between groups in Patients' Endorsement of a Biopsychosocial Model of Pain/Persistent Somatic Symptoms (PEB) score | T1(before randomization), T2 (week 6, mid-treatment), T3 (primary endpoint, 12 weeks), T4 (3-month follow-up), T5 (1-year follow-up), T6 (2-year follow-up)
  The participants' bio-psycho-social understanding of their symptoms will we measured using the 11 item PEB questionnaire. The PEB is developed to measure patients' specific beliefs regarding pain. The scale has been adjusted to include a broader spectrum of physical symptoms relevant to functional somatic disorder instead of focusing on pain alone. Items are rated on a 4-point Likert scale resulting in a total score ranging from 11-44 with higher scores indicating a better bio-psycho-social understanding.
Mean difference between groups in Numeric Rating Scale (NRS) on symptom intensity and symptom interference | T0 (baseline, before assessment), T1(before randomization), T2 (week 6, mid-treatment), T3 (primary endpoint, 12 weeks), T4 (3-month follow-up), T5 (1-year follow-up), T6 (2-year follow-up)
  Symptom intensity and symptom interference is measured on a NRS ranging 0 to 10 on 2 items. This results in scores ranging from 0 to 20 with higher scores meaning worse symptoms.
Mean difference between groups in Numeric Rating Scale (NRS) on pain intensity | T0 (baseline, before assessment), T1(before randomization), T2 (week 6, mid-treatment), T3 (primary endpoint, 12 weeks), T4 (3-month follow-up), T5 (1-year follow-up), T6 (2-year follow-up)
  Pain intensity is measured on a NRS ranging 0 to 10 on 1 item. A higher score indicates higher pain intensity.
Mean difference between groups in Brief-Illness Perception Questionnaire (b-IPQ) | T0 (baseline, before assessment), T1(before randomization), T2 (week 6, mid-treatment), T3 (primary endpoint, 12 weeks), T4 (3-month follow-up), T5 (1-year follow-up), T6 (2-year follow-up)
  Illness perception is measured using b-IPQ, containing 8 items each scored on a 11-point scale from 0 to 10. This results in a total score ranging from 0 to 80 with higher scores indicating more negative illness perception.
Mean difference between groups in Behavioural Responses to Illness Questionnaire (BRIQ) | T0 (baseline, before assessment), T1(before randomization), T2 (week 6, mid-treatment), T3 (primary endpoint, 12 weeks), T4 (3-month follow-up), T5 (1-year follow-up), T6 (2-year follow-up)
  Illness behaviour is measured using the BRIQ containing 13 items scored on a 5 point Likert scale. This results in a total score from 13 to 65 with higher scores indicating more negative illness behaviour.
Mean difference between groups in clinician-rated Clinical Global Improvement Scale (CGI) score | T3 (primary endpoint, 12 weeks)
  Clinician-rated overall health improvement measured by the 5-point CGI. Clinicians are asked to rate the patient's general health as "much worse", "worse", "unchanged", "better" or "much better" in response to the question: "How do you consider your patient's health status now compared with when the patient first came to the clinic?"
Mean difference between groups in diagnosis based on a clinical diagnostic reassessment | T3 (primary endpoint, 12 weeks)
  Doctors will evaluate if the diagnostic criteria for multisystem functional somatic disorder, operationalized using the criteria for multiorgan bodily distress syndrome.

OTHER OUTCOMES:
Mean score on a patient-rated Numeric Rating Scale (NRS) regarding expected effect of study drug | T1(before randomization)
  For participants in the study drug trial, expected effect of the study drug on their overall wellbeing will be measured using a 11-point NRS ranging from 0 to 10 with higher scores meaning higher expectations to the effect of the study drug.
Mean score on a clinician-rated Numeric Rating Scale (NRS) regarding expected effect of study drug | T1(before randomization)
  Clinicians will be asked to evaluate their expectations for the effect of the study drug on the overall health improvement for participants in the study drug trial. This will be measured using an 11-point NRS ranging from 0 to 10 with higher scores meaning higher expectations to the effect of the study drug.
Mean score on Spiritual Needs Questionnaire (SNQ) | T1(before randomization)
  The existential needs of the patient is measured using the SNQ. Participants will rate 20 items representing their spiritual needs on four domains: Religious needs, existential needs, inner peace needs, and generativity needs. Items are rated from 0 (No) to 3 (Very big). This results in a total score ranging from 0 to 60 with higher scores indicating higher spiritual needs. The participants will additionally be asked to rate if they felt like such needs were adressed in the assessment, if they felt like such a focus was missing from the assessment, if they found such a focus to be relevant, if they felt like a doctor should adress such needs and if they found that others (presented in a list) would be more relevant to adress such needs with.
Mean difference between groups on the Credibility/Expectancy Questionnaire (CEQ) | T2 (week 6, mid-treatment)
  Patients expectations of treatment effects (both PE and study drug treatment) will be measured by the CEQ containing 6 items rated from 1 to 10 resulting in a total score from 6 to 60 with higher scores indicating higher confidence in the treatment offered.
Mean score on Inventory for the Assessment of Negative Effects of Psychotherapy (INEP) | T3 (primary endpoint, 12 weeks)
  The Inventory for the assessment of Negative Effects of Psychotherapy (INEP) contains 21 items covering e.g. relationships problems, dependence on the therapist, and financial worries. Respondents are asked to indicate on a 4-point scale to what extent they agree or disagree with these statements. Other items are answered on a 3-point scale, e.g. "I feel…": "better", "unchanged/not applicable" or "worse".
  Negative effects of psychological treatment is measured by the INEP with 21 items with some items rated on a 4 point scale and others on a 3 points scale.
  Higher scores indicate experience of more negative effects.
Mean score on Working Alliance Inventory-Short revised (WAI-SR) | T2 (week 6, mid-treatment) and T3 (primary endpoint, 12 weeks)
  Patients and clinicians relationship will be measured by the 12 item WAI-SR questionnaire. Items will be scored on a 7 point scale with higher scores indicating a better working alliance.
European Quality of Life - 5 dimensions (EQ-D5) | T1(before randomization), T2 (week 6, mid-treatment), T3 (primary end-point, 12 weeks), T5 (1-year follow-up), T6 (2-year follow-up)
  Data on health economic measures will be calculated by use of the EQ-D5 quality of life measure.
Mean difference between groups in participants' recollection of the content of patient education (PE) program | T3 (primary endpoint, 12 weeks)
  For participants in the PE intervention, six questions on participant's recollection of the content of the PE program will be scored on a three point scale.
Mean difference between groups on the Sources of Meaning and Meaning in Life, Danish version) (SoMe-Da) score | T1(before randomization), T3 (primary endpoint, 12 weeks), T4 (3-month follow-up)
  Experience of meaning in life and crisis is measured using the 10 item SoMe-Da. Items are rated on a 6 point scale with higher scores indicating more experience of meaning in life.
Mean score on the Experience of Service Questionnaire (ESQ) | T3 (primary endpoint, 12 weeks)
  Participants' satisfaction with the interventions will be measured using the ESQ. It is a 15-item questionnaire made up of 12 statements (about facilities, staff, how well the patient was treated, confidence in staff, and overall satisfaction with the service) and three additional questions which invite free text responses: 'What was really good about your care?'; 'Was there anything you didn't like or anything that needs improving?'; and 'Is there anything else you want to tell us about the service you received?'. The 12 statements are rated on a Likert scale to determine the level of agreement (certainly true, scoring 1; partly true, scoring 0; not true, scoring -1, and don't know, not scored); scores range from 12 (very satisfied) to -12 (very dissatisfied).
Change in blood pressure following study drug treatment | Before study drug treatment initiation, at visits at the clinic in week 3, week 7 or 8 and week 12.
  As hypertension is a known side effect to duloxetin, blood pressure will be meassured before and during study drug treatment and this measure will be reported.
Concentration of duloxetine in serum | T3 (primary endpoint, 12 weeks)
  A blood test will be taken in order to measure serum duloxetine in all participants in the study drug trial to evaluate compliance. The results will be analyzed at the end of the trial and remain blinded from all study personel throughout data analysis.
Differences between groups in concentration of biomarkers in blood samples | Week 3 and week 12
  2 glasses of 10 ml will be drawn for coagulation blood and 2 glasses of 10 ml for EDTA-blood to investigate biomarkers for functional disorder. Participants will have been fasting for 12 hours or more when samples are collected.
  Analysis will include concentration of proinflammatory cytokines and such as IL-1RA, IL-6, and IL-8 and chemokines such as CCL17, CCL22, CXCL9, and CXCL11. Additionally, biomarkers indicating an over-activated kynurenine pathway and C-reactive protein (CRP) and the specialized pro-resolving lipid mediators (SPM) will be meassured. Neuroendocrine dysfunction will be investigated by meassuring the corticotropin-releasing hormone (CRH), the monoamines serotonin, noradrenaline, and dopamine and their metabolites 5-HIAA, DOPAC, and HVA, as well as the neuropeptide Substance P and tumor necrosis factor (TNF).
Diary of diet and medication | 3 days prior to collection of biological material in week 3 and week 12
  Participants will be asked to write a diary of their diet and medication three days prior to the collection of biological samples
Differences between groups in biomarkers in feces samples | Week 3 and week 12
  The participant will bring feces samples from home for investigation of the mikrobiota. This will be done exploratively through laboratory analysis of different signaling molecules such as metabolites, neuromodulators, neuropeptides, and neurotransmitters.

CONTACTS AND LOCATIONS:
Overall Officials: Lise K Gormsen, MD, PhD, Principal Investigator — Department of Funtional disorders, Aarhus University Hospital
Locations (1):
- Research Cinic for Functional Disorders, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Before and during the study the Study protocol, statistical analysis plan and inform consent form can be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 2024-2027
Access Criteria: independent researcher in the area.

REFERENCES:
- [Background] Burton C, Fink P, Henningsen P, Lowe B, Rief W; EURONET-SOMA Group. Functional somatic disorders: discussion paper for a new common classification for research and clinical use. BMC Med. 2020 Mar 3;18(1):34. doi: 10.1186/s12916-020-1505-4. PMID 32122350
- [Background] Roenneberg C, Sattel H, Schaefert R, Henningsen P, Hausteiner-Wiehle C. Functional Somatic Symptoms. Dtsch Arztebl Int. 2019 Aug 9;116(33-34):553-560. doi: 10.3238/arztebl.2019.0553. PMID 31554544
- [Background] Henningsen P, Zipfel S, Sattel H, Creed F. Management of Functional Somatic Syndromes and Bodily Distress. Psychother Psychosom. 2018;87(1):12-31. doi: 10.1159/000484413. Epub 2018 Jan 6. PMID 29306954
- [Background] Petersen MW, Schroder A, Jorgensen T, Ornbol E, Dantoft TM, Eliasen M, Carstensen TW, Falgaard Eplov L, Fink P. Prevalence of functional somatic syndromes and bodily distress syndrome in the Danish population: the DanFunD study. Scand J Public Health. 2020 Jul;48(5):567-576. doi: 10.1177/1403494819868592. Epub 2019 Aug 14. PMID 31409218
- [Background] Fink P, Schroder A. One single diagnosis, bodily distress syndrome, succeeded to capture 10 diagnostic categories of functional somatic syndromes and somatoform disorders. J Psychosom Res. 2010 May;68(5):415-26. doi: 10.1016/j.jpsychores.2010.02.004. PMID 20403500
- [Background] Hauser W, Hausteiner-Wiehle C, Henningsen P, Brahler E, Schmalbach B, Wolfe F. Prevalence and overlap of somatic symptom disorder, bodily distress syndrome and fibromyalgia syndrome in the German general population: A cross sectional study. J Psychosom Res. 2020 Jun;133:110111. doi: 10.1016/j.jpsychores.2020.110111. Epub 2020 Apr 11. PMID 32305723
- [Background] Fink P, Toft T, Hansen MS, Ornbol E, Olesen F. Symptoms and syndromes of bodily distress: an exploratory study of 978 internal medical, neurological, and primary care patients. Psychosom Med. 2007 Jan;69(1):30-9. doi: 10.1097/PSY.0b013e31802e46eb. PMID 17244846
- [Background] Budtz-Lilly A, Vestergaard M, Fink P, Carlsen AH, Rosendal M. Patient characteristics and frequency of bodily distress syndrome in primary care: a cross-sectional study. Br J Gen Pract. 2015 Sep;65(638):e617-23. doi: 10.3399/bjgp15X686545. PMID 26324499
- [Background] Rask MT, Rosendal M, Fenger-Gron M, Bro F, Ornbol E, Fink P. Sick leave and work disability in primary care patients with recent-onset multiple medically unexplained symptoms and persistent somatoform disorders: a 10-year follow-up of the FIP study. Gen Hosp Psychiatry. 2015 Jan-Feb;37(1):53-9. doi: 10.1016/j.genhosppsych.2014.10.007. Epub 2014 Oct 22. PMID 25456975
- [Background] Schroder A, Ornbol E, Jensen JS, Sharpe M, Fink P. Long-term economic evaluation of cognitive-behavioural group treatment versus enhanced usual care for functional somatic syndromes. J Psychosom Res. 2017 Mar;94:73-81. doi: 10.1016/j.jpsychores.2017.01.005. Epub 2017 Jan 10. PMID 28183406
- [Background] van Dessel N, den Boeft M, van der Wouden JC, Kleinstauber M, Leone SS, Terluin B, Numans ME, van der Horst HE, van Marwijk H. Non-pharmacological interventions for somatoform disorders and medically unexplained physical symptoms (MUPS) in adults. Cochrane Database Syst Rev. 2014 Nov 1;2014(11):CD011142. doi: 10.1002/14651858.CD011142.pub2. PMID 25362239
- [Background] Schroder A, Rehfeld E, Ornbol E, Sharpe M, Licht RW, Fink P. Cognitive-behavioural group treatment for a range of functional somatic syndromes: randomised trial. Br J Psychiatry. 2012 Jun;200(6):499-507. doi: 10.1192/bjp.bp.111.098681. Epub 2012 Apr 26. PMID 22539780
- [Background] Fjorback LO, Arendt M, Ornbol E, Walach H, Rehfeld E, Schroder A, Fink P. Mindfulness therapy for somatization disorder and functional somatic syndromes: randomized trial with one-year follow-up. J Psychosom Res. 2013 Jan;74(1):31-40. doi: 10.1016/j.jpsychores.2012.09.006. Epub 2012 Oct 1. PMID 23272986
- [Background] Agger JL, Schroder A, Gormsen LK, Jensen JS, Jensen TS, Fink PK. Imipramine versus placebo for multiple functional somatic syndromes (STreSS-3): a double-blind, randomised study. Lancet Psychiatry. 2017 May;4(5):378-388. doi: 10.1016/S2215-0366(17)30126-8. Epub 2017 Apr 10. PMID 28408193
- [Background] Pedersen HF, Agger JL, Frostholm L, Jensen JS, Ornbol E, Fink P, Schroder A. Acceptance and Commitment group Therapy for patients with multiple functional somatic syndromes: a three-armed trial comparing ACT in a brief and extended version with enhanced care. Psychol Med. 2019 Apr;49(6):1005-1014. doi: 10.1017/S0033291718001666. Epub 2018 Jun 26. PMID 29941062
- [Background] Hauser W, Ablin J, Perrot S, Fitzcharles MA. Management of fibromyalgia: practical guides from recent evidence-based guidelines. Pol Arch Intern Med. 2017 Jan 4;127(1):47-56. doi: 10.20452/pamw.3877. Epub 2017 Jan 4. PMID 28075425
- [Background] Carville S, Constanti M, Kosky N, Stannard C, Wilkinson C; Guideline Committee. Chronic pain (primary and secondary) in over 16s: summary of NICE guidance. BMJ. 2021 Apr 21;373:n895. doi: 10.1136/bmj.n895. No abstract available. PMID 33883123
- [Background] Clauw DJ. Fibromyalgia: a clinical review. JAMA. 2014 Apr 16;311(15):1547-55. doi: 10.1001/jama.2014.3266. PMID 24737367
- [Background] Ford AC, Lacy BE, Talley NJ. Irritable Bowel Syndrome. N Engl J Med. 2017 Jun 29;376(26):2566-2578. doi: 10.1056/NEJMra1607547. No abstract available. PMID 28657875
- [Background] Kleinstauber M, Witthoft M, Hiller W. Efficacy of short-term psychotherapy for multiple medically unexplained physical symptoms: a meta-analysis. Clin Psychol Rev. 2011 Feb;31(1):146-60. doi: 10.1016/j.cpr.2010.09.001. Epub 2010 Sep 16. PMID 20920834
- [Background] Christensen SS, Frostholm L, Ornbol E, Schroder A. Changes in illness perceptions mediated the effect of cognitive behavioural therapy in severe functional somatic syndromes. J Psychosom Res. 2015 Apr;78(4):363-70. doi: 10.1016/j.jpsychores.2014.12.005. Epub 2014 Dec 13. PMID 25541119
- [Background] Gruman J, Rovner MH, French ME, Jeffress D, Sofaer S, Shaller D, Prager DJ. From patient education to patient engagement: implications for the field of patient education. Patient Educ Couns. 2010 Mar;78(3):350-6. doi: 10.1016/j.pec.2010.02.002. Epub 2010 Mar 3. PMID 20202780
- [Background] Hoving C, Visser A, Mullen PD, van den Borne B. A history of patient education by health professionals in Europe and North America: from authority to shared decision making education. Patient Educ Couns. 2010 Mar;78(3):275-81. doi: 10.1016/j.pec.2010.01.015. Epub 2010 Mar 1. PMID 20189746
- [Background] Frolund Pedersen H, Holsting A, Frostholm L, Rask C, Jensen JS, Hoeg MD, Schroder A. "Understand your illness and your needs": Assessment-informed patient education for people with multiple functional somatic syndromes. Patient Educ Couns. 2019 Sep;102(9):1662-1671. doi: 10.1016/j.pec.2019.04.016. Epub 2019 Apr 17. PMID 31023608
- [Background] Kleinstauber M, Witthoft M, Steffanowski A, van Marwijk H, Hiller W, Lambert MJ. Pharmacological interventions for somatoform disorders in adults. Cochrane Database Syst Rev. 2014 Nov 7;2014(11):CD010628. doi: 10.1002/14651858.CD010628.pub2. PMID 25379990
- [Background] Welsch P, Uceyler N, Klose P, Walitt B, Hauser W. Serotonin and noradrenaline reuptake inhibitors (SNRIs) for fibromyalgia. Cochrane Database Syst Rev. 2018 Feb 28;2(2):CD010292. doi: 10.1002/14651858.CD010292.pub2. PMID 29489029
- [Background] Hirase T, Hirase J, Ling J, Kuo PH, Hernandez GA, Giwa K, Marco R. Duloxetine for the Treatment of Chronic Low Back Pain: A Systematic Review of Randomized Placebo-Controlled Trials. Cureus. 2021 May 22;13(5):e15169. doi: 10.7759/cureus.15169. PMID 34046287
- [Background] Rodrigues-Amorim D, Olivares JM, Spuch C, Rivera-Baltanas T. A Systematic Review of Efficacy, Safety, and Tolerability of Duloxetine. Front Psychiatry. 2020 Oct 23;11:554899. doi: 10.3389/fpsyt.2020.554899. eCollection 2020. PMID 33192668
- [Background] Rosenblat JD, Kakar R, McIntyre RS. The Cognitive Effects of Antidepressants in Major Depressive Disorder: A Systematic Review and Meta-Analysis of Randomized Clinical Trials. Int J Neuropsychopharmacol. 2015 Jul 25;19(2):pyv082. doi: 10.1093/ijnp/pyv082. PMID 26209859
- [Background] Barber AJ, Tischler VA, Healy E. Consumer satisfaction and child behaviour problems in child and adolescent mental health services. J Child Health Care. 2006 Mar;10(1):9-21. doi: 10.1177/1367493506060200. PMID 16464930
- [Background] Fink P. Syndromes of bodily distress or functional somatic syndromes - Where are we heading. Lecture on the occasion of receiving the Alison Creed award 2017. J Psychosom Res. 2017 Jun;97:127-130. doi: 10.1016/j.jpsychores.2017.04.012. Epub 2017 Apr 25. No abstract available. PMID 28606492
- [Background] Petersen MW, Schroder A, Jorgensen T, Ornbol E, Meinertz Dantoft T, Eliasen M, Benros ME, Fink P. Irritable bowel, chronic widespread pain, chronic fatigue and related syndromes are prevalent and highly overlapping in the general population: DanFunD. Sci Rep. 2020 Feb 24;10(1):3273. doi: 10.1038/s41598-020-60318-6. PMID 32094442
- [Background] Kallesoe KH, Schroder A, Jensen JS, Wicksell RK, Rask CU. Group-based Acceptance and Commitment Therapy (AHEAD) for adolescents with multiple functional somatic syndromes: A randomised trial. JCPP Adv. 2021 Dec 8;1(4):e12047. doi: 10.1002/jcv2.12047. eCollection 2021 Dec. PMID 37431406
- [Background] Wallace DJ, Linker-Israeli M, Hallegua D, Silverman S, Silver D, Weisman MH. Cytokines play an aetiopathogenetic role in fibromyalgia: a hypothesis and pilot study. Rheumatology (Oxford). 2001 Jul;40(7):743-9. doi: 10.1093/rheumatology/40.7.743. PMID 11477278
- [Background] Vaeroy H, Helle R, Forre O, Kass E, Terenius L. Elevated CSF levels of substance P and high incidence of Raynaud phenomenon in patients with fibromyalgia: new features for diagnosis. Pain. 1988 Jan;32(1):21-26. doi: 10.1016/0304-3959(88)90019-X. PMID 2448729
- [Background] Tsilioni I, Russell IJ, Stewart JM, Gleason RM, Theoharides TC. Neuropeptides CRH, SP, HK-1, and Inflammatory Cytokines IL-6 and TNF Are Increased in Serum of Patients with Fibromyalgia Syndrome, Implicating Mast Cells. J Pharmacol Exp Ther. 2016 Mar;356(3):664-72. doi: 10.1124/jpet.115.230060. Epub 2016 Jan 13. PMID 26763911
- [Background] Thompson T, Gallop K, Correll CU, Carvalho AF, Veronese N, Wright E, Stubbs B. Pain perception in Parkinson's disease: A systematic review and meta-analysis of experimental studies. Ageing Res Rev. 2017 May;35:74-86. doi: 10.1016/j.arr.2017.01.005. Epub 2017 Feb 4. PMID 28179128
- [Background] Rodriguez-Pinto I, Agmon-Levin N, Howard A, Shoenfeld Y. Fibromyalgia and cytokines. Immunol Lett. 2014 Oct;161(2):200-3. doi: 10.1016/j.imlet.2014.01.009. Epub 2014 Jan 23. PMID 24462815
- [Background] Papadopoulos AS, Cleare AJ. Hypothalamic-pituitary-adrenal axis dysfunction in chronic fatigue syndrome. Nat Rev Endocrinol. 2011 Sep 27;8(1):22-32. doi: 10.1038/nrendo.2011.153. PMID 21946893
- [Background] Neeck G, Riedel W. Neuromediator and hormonal perturbations in fibromyalgia syndrome: results of chronic stress? Baillieres Clin Rheumatol. 1994 Nov;8(4):763-75. doi: 10.1016/s0950-3579(05)80047-0. PMID 7850879
- [Background] Liu L, Wu Q, Chen Y, Ren H, Zhang Q, Yang H, Zhang W, Ding T, Wang S, Zhang Y, Liu Y, Sun J. Gut microbiota in chronic pain: Novel insights into mechanisms and promising therapeutic strategies. Int Immunopharmacol. 2023 Feb;115:109685. doi: 10.1016/j.intimp.2023.109685. Epub 2023 Jan 24. PMID 37278059
- [Background] Hagelberg N, Jaaskelainen SK, Martikainen IK, Mansikka H, Forssell H, Scheinin H, Hietala J, Pertovaara A. Striatal dopamine D2 receptors in modulation of pain in humans: a review. Eur J Pharmacol. 2004 Oct 1;500(1-3):187-92. doi: 10.1016/j.ejphar.2004.07.024. PMID 15464032
- [Background] Groven N, Reitan SK, Fors EA, Guzey IC. Kynurenine metabolites and ratios differ between Chronic Fatigue Syndrome, Fibromyalgia, and healthy controls. Psychoneuroendocrinology. 2021 Sep;131:105287. doi: 10.1016/j.psyneuen.2021.105287. Epub 2021 May 27. PMID 34090138
- [Background] Demitrack MA, Dale JK, Straus SE, Laue L, Listwak SJ, Kruesi MJ, Chrousos GP, Gold PW. Evidence for impaired activation of the hypothalamic-pituitary-adrenal axis in patients with chronic fatigue syndrome. J Clin Endocrinol Metab. 1991 Dec;73(6):1224-34. doi: 10.1210/jcem-73-6-1224. PMID 1659582
- [Background] Cleare AJ. The neuroendocrinology of chronic fatigue syndrome. Endocr Rev. 2003 Apr;24(2):236-52. doi: 10.1210/er.2002-0014. PMID 12700181
- [Background] Amin OA, Abouzeid SM, Ali SA, Amin BA, Alswat KA. Clinical association of vitamin D and serotonin levels among patients with fibromyalgia syndrome. Neuropsychiatr Dis Treat. 2019 May 27;15:1421-1426. doi: 10.2147/NDT.S198434. eCollection 2019. PMID 31239680
- [Derived] Jespersen CP, Pedersen HF, Kleinstauber M, Fink P, Wellnitz KB, Ornbol E, Schroder A, Agger JL, Vase L, Finnerup NB, Gormsen LK. Efficacy of patient education and duloxetine, alone and in combination, for patients with multisystem functional somatic disorder: Study protocol for the EDULOX trial. Contemp Clin Trials. 2024 Jun;141:107524. doi: 10.1016/j.cct.2024.107524. Epub 2024 Apr 9. PMID 38604496
- See also: US Natl Inst Health. Current medication information for benztropine mesylate, A.a. Accessed August 2020. — https://dailymed.nlm.nih.gov/dailymed/index.cfm